CLINICAL TRIAL: NCT05726162
Title: Effects of Biofeedback-based Music Program Using a Smart Device Application on Perioperative Sleep Quality in Patients Undergoing Breast Cancer Surgery: an Open-labeled Randomized Controlled Study
Brief Title: Effects of Biofeedback-based Music Program Using a Smart Device Application on Perioperative Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Biofeedback_based_music
Record Dates: First submitted 2023-01-30; First posted 2023-02-13 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients sleep as usual with noise-canceling earplugs
  Interventions: Other: Control
- Biofeedback-based music (Experimental): Patient is provided with a biofeedback-based music program using a smart device application for sleep.
  Interventions: Device: biofeedback-based music program

INTERVENTIONS:
Device: biofeedback-based music program — The investigators will provide biofeedback-based music, which incorporates the patient's respiratory information. In a biofeedback-based music group, the patient performs an active respiratory intervention session, which induces a slow breathing pattern. If breathing has been slow enough, the automatic mode is activated to provide music based on patient's own breathing pattern. It automatically will be terminated 30 minutes after intervention.
  Arms: Biofeedback-based music
Other: Control — The investigators will provide noise-canceling earplugs to minimize bias from noise in the ward.
  Arms: Control

SUMMARY:
The purpose of this study is to investigate whether the effects of biofeedback-based music programs using a smart device application can improve perioperative sleep quality in patients undergoing breast cancer surgery.

DETAILED DESCRIPTION:
In a biofeedback-based music group, the patient performs an active respiratory intervention session, which induces a slow breathing pattern. If breathing has been slow enough, the automatic mode is activated to provide music based on the patient's own breathing pattern. The investigators will provide biofeedback-based music, which incorporates the patient's respiratory information, while no intervention will be performed in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective breast cancer surgery

Exclusion Criteria:

* Patients' refusal
* Day surgery or urgent surgery
* BMI ≥35
* Neurocognitive impairment, hearing disorder (ex : (dementia, impaired cognitive dysfunction, cerebral infarction, transient cerebral ischemic attack))
* Patients with psychiatric diseases, psychological drug intake
* Pre-existing conditions associated with sleep disorders or drug intake related to sleep

Ages: 19 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The Richards-Campbell Sleep Questionnaire on the day of the surgery | The daytime after the surgery (POD1)
  sleep quality questionnaires that are most commonly used in the ICU setting, RCSQ 1-5 (0-100), Average RCSQ (0-100), higher scores mean a better outcome

SECONDARY OUTCOMES:
The Richards-Campbell Sleep Questionnaire on the day before the surgery | on the day of the surgery before surgery
  sleep quality questionnaires that are most commonly used in the ICU setting, RCSQ 1-5 (0-100), Average RCSQ (0-100), higher scores mean a better outcome
Pittsburgh Sleep Quality Index | on the day before the surgery
  A self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. C1-7 (0-3), total (0-21), higher scores mean a worse outcome
Quality of recovery score 15 (QoR 15) | on the day before the surgery
  Korean version of quality of recovery-15 (0-150), higher scores mean a better outcome
Hospital Anxiety and Depression scale | on the day before the surgery
  Method to measure anxiety and depression in a general medical population of patient, total (0-42), K-HADS depression subscale(0-21), K-HADS anxiety (0-21), higher scores mean a worse outcome
The Richards-Campbell Sleep Questionnaire (baseline, usual patients' pattern) | on the day before the surgery
  sleep quality questionnaires that are most commonly used in the ICU setting, RCSQ 1-5 (0-100), Average RCSQ (0-100), higher scores mean a better outcome
Quality of recovery score 15 (QoR 15) | after the surgery (POD1; Postoperative 24 hours)
  Korean version of quality of recovery-15 (0-150), higher scores mean a better outcome
Postoperative Pain | after the surgery (POD1; Postoperative 24 hours)
  NRS score (0-11) of pain, higher scores mean a worse outcome
The incidence of postoperative nausea and vomiting | after the surgery (POD1; Postoperative 24 hours)
  Postoperative nausea and vomiting
Postoperative opioid consumption | after the surgery (POD1; Postoperative 24 hours)
  Postoperative opioid requirement
Analgesics requirement | after the surgery (POD1; Postoperative 24 hours)
  Analgesics other than opioid requirement
Total sleep time (hours) | The daytime after the surgery (POD1)
  Duration of sleep
Time to fall asleep (minutes) | The daytime after the surgery (POD1)
  The time to sleep from intervention
Sleep quality (0-100) | The daytime after the surgery (POD1)
  VAS score for sleep quality (0-100), higher scores mean a better outcome
Sleep disturbance | The daytime after the surgery (POD1)
  Awakened from sleep (yes/no)
The reasons of sleep disturbance | The daytime after the surgery (POD1)
  Ask the patients who answered "yes" to the question of whether there was a disturbance during sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Seohee Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea